CLINICAL TRIAL: NCT01508000
Title: Randomized Phase II Trial Evaluating the Efficacy of FOLFOX Alone, FOLFOX Plus Bevacizumab and FOLFOX Plus Panitumumab as Perioperative Treatment in Patients With Resectable Liver Metastases From Wild Type KRAS/NRAS Colorectal Cancer
Brief Title: Efficacy of FOLFOX Alone, FOLFOX Plus Bevacizumab and FOLFOX Plus Panitumumab in Patients With Resectable Liver Metastases
Acronym: BOS2
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Low or poor accrual
Sponsor: European Organisation for Research and Treatment of Cancer - EORTC (Network)
Collaborators: Amgen (Industry); Roche Pharma AG (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EORTC-40091; 2010-019238-29 (EudraCT Number)
Record Dates: First submitted 2012-01-09; First posted 2012-01-11 (Estimated); Last update posted 2016-10-12 (Estimated); Status verified 2016-10

CONDITIONS: Colorectal Cancer Metastatic; Liver Metastases; KRAS Wild Type Colorectal Cancer
Keywords: Liver metastases; Colorectal Cancer; KRAS wild type; FOLFOX; Bevacizumab; Panitumumab; Randomized; Phase II; Perioperative treatment; Adjuvant; Neo-adjuvant; Surgery; Progression Free Survival
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Folfox protocol; Drug Therapy; Bevacizumab; Panitumumab; Surgical Procedures, Operative

ARMS (3):
- Arm A: modified FOLFOX6 and Surgery (Active Comparator): 6 cycles before and 6 cycles after surgery consisting in:
  Hour 0: Oxaliplatin 85 mg/m² IV 2-h infusion
  Hour 0: Folinic Acid 400 mg/m² (DL form) or 200 mg/m2 (L form) IV 2-h infusion
  Hour 2: 5-FU 400 mg/m² IV bolus over 2-4 minutes
  Hour 2: 5-FU 2400 mg/m² given as a continuous infusion over 46h.
  On day 1 of a 14 day cycle
  Interventions: Drug: FOLFOX6; Procedure: Surgery
- Arm B: modified FOLFOX6 + Bevacizumab and Surgery (Experimental): 6 cycles before and 6 cycles after surgery consisting in:
  Hour 0: Oxaliplatin 85 mg/m2 2-h infusion
  Hour 0: Folinic Acid 400 mg/m2 (DL form) or 200 mg/m2 (L form) 2-h infusion
  Hour 2 (before 5-FU bolus): Bevacizumab 5 mg/kg IV over 90 minutes infusion*.
  Hour 3.5: 5-FU bolus 400 mg/m2 IV bolus over 2-4 minutes
  Hour 3.5: 5-FU 2400 mg/m² given as a continuous infusion over 46h.
  On day 1 of a 14 day cycle
  Interventions: Drug: FOLFOX6; Biological: Bevacizumab; Procedure: Surgery
- Arm C: modified FOLFOX6 + Panitumumab and Surgery (Experimental): Experimental: Arm B: modified FOLFOX6 + Bevacizumab and Surgery
  6 cycles before and 6 cycles after surgery consisting in:
  Hour - 1 (pre chemotherapy): Panitumumab 6 mg/kg IV over 60 minutes (≤ 1000 mg) or 90 minutes (> 1000 mg) +/- 15 min. infusion*.
  Hour 0: Oxaliplatin 85 mg/m² IV 2-h infusion
  Hour 0: Folinic Acid 400 mg/m² (DL form) or 200 mg/m2 (L form) IV 2-h infusion
  Hour 2: 5-FU 400 mg/m² IV bolus over 2-4 minutes
  Hour 2: 5-FU 2400 mg/m² given as a continuous infusion over 46h.
  On day 1 of a 14 day cycle
  Interventions: Drug: FOLFOX6; Biological: Panitumumab; Procedure: Surgery

INTERVENTIONS:
Drug: FOLFOX6 — 5-FU, folinic acid, oxaliplatin
  Other Names: Chemotherapy
Biological: Bevacizumab — Targeted therapy
  Other Names: Avastin
  Arms: Arm B: modified FOLFOX6 + Bevacizumab and Surgery
Biological: Panitumumab — Targeted therapy
  Other Names: Vectibix
  Arms: Arm C: modified FOLFOX6 + Panitumumab and Surgery
Procedure: Surgery

SUMMARY:
Patients presenting with multiple innumerable liver metastases will probably never come to resection, however, for all others, including patients with numerous multiple metastases or large metastases,resection should be considered after limited chemotherapy.

There is consensus for a backbone chemotherapy consisting of fluoropyrimidine + oxaliplatin. FOLFOX was used in the previous EORTC study and is again recommended.

The addition of targeted agents to standard chemotherapy in the perioperative strategy for mCRC might increase the ORR and R0 resectability, without significant increase in toxicity, therefore translating to a better outcome.

It was therefore decided to design an open label, randomized, multi-center, 3-arm late phase II study.

Arm A: (standard) mFOLFOX6 + Surgery Arm B: (experimental) mFOLFOX6 + Bevacizumab + Surgery Arm C: (experimental) mFOLFOX6 + Panitumumab + Surgery

ELIGIBILITY:
Inclusion Criteria:

* Histologically proven CRC with 1 to 8 metachronous or synchronous liver metastases considered to be completely resectable.
* Primary tumor (or liver metastasis) of CRC must be KRAS and NRAS status "wild type".
* Patients must have undergone complete resection (R0) of the primary tumor at least 4 weeks before randomization. Or for patients with synchronous metastases the primary tumor can be resected (R0) at the same time as the liver metastases if: the patient has a non-obstructive primary tumor and is able to receive preoperative chemotherapy (3-4 months) before surgery.
* Measurable hepatic disease by RECIST version 1.1.
* Patients must be 18 years old or older.
* A WHO performance status of 0 or 1. Radiotherapy alone is allowed if given pre or post protocol treatment.
* Previous adjuvant chemotherapy for primary CRC is allowed if completed at least 12 months before inclusion in this study.
* All the following tests should be done within 4 weeks prior to randomization:
* Absolute neutrophil count ≥ 1.5 x 109/L, platelets ≥ 100 x 109/L, hemoglobin ≥ 9 g/dL and white blood cell count (WBC) ≥ 3 x 109/L.
* Serum creatinine ≤ 1.5 times the upper limit of normal (ULN) (to exclude severe renal impairment); no significant proteinuria (urine protein < 1g/24 hours urine collection) OR urine protein/creatinine ratio < 1.0 OR 1+ proteinuria on urine dipstick.
* Absence of major hepatic insufficiency (bilirubin ≤ 1.5 x ULN and aspartate aminotransferase (ASAT) and alanine aminotransferase (ALAT) ≤ 5 x ULN).
* Magnesium ≥ lower limit of normal (LLN)
* Patients with a buffer range from the normal values of +/- 5% for hematology and +/- 10% for biochemistry are acceptable. This will not apply for Renal Function, including Creatinine.
* Women of child bearing potential (WOCBP) must have a negative serum (or urine) pregnancy test within 14 days prior to the first dose of study treatment.
* Patients of childbearing / reproductive potential should use adequate birth control measures, as defined by the investigator, during the study treatment period and for at least 6 months after the last study treatment. A highly effective method of birth control is defined as those which result in low failure rate (i.e. less than 1% per year) when used consistently and correctly.
* Female subjects who are breast feeding should discontinue nursing prior to the first dose of study treatment and until 6 months after the last study treatment.
* Before patient registration/randomization, written informed consent must be given according to ICH/GCP, and national/local regulations.

Exclusion Criteria:

* Evidence of extra-hepatic metastasis (of CRC).
* Previous chemotherapy for metastatic disease or surgical treatment (e.g. surgical resection or radiofrequency ablation) for liver metastasis.
* Previous exposure to EGFR or VEGF/VEGFR targeting therapy within the last 12 months.
* Major surgical procedure, open biopsy, or significant traumatic injury within 4 weeks prior to randomization.
* Regular use of aspirin or other non-steroidal anti-inflammatory drugs (NSAIDs).
* Bleeding diathesis (e.g. hemoptysis of ≥ 1/2 teaspoon or 2.5mL), coagulopathy, or need for administration of full-dose anti-coagulant(s).
* Clinically significant cardiovascular disease, including: uncontrolled hypertension, New York Heart Association (NYHA) class II-IV heart failure, myocardial infarction or unstable angina pectoris, cerebrovascular accident or transient ischemic attack within the past 12 months, peripheral vascular disease ≥ grade 2, serious cardiac arrhythmia requiring medication and other clinically significant cardiovascular disease.
* Peripheral neuropathy > grade 1 (Common Terminology Criteria for Adverse Events, v4.0) serious wound complications, ulcers, or bone fractures.
* Symptomatic diverticulitis or active or uncontrolled gastroduodenal ulceration.
* History or evidence of interstitial lung disease (e.g. pneumonitis, pulmonary fibrosis)
* Significant disease that, in the investigator's opinion, would exclude the patient from the study. Including known allergy or any other adverse reaction to any of the study drugs (including any of the excipients) or to any related compound, including hypersensitivity to Chinese hamster ovary (CHO) cell products or other recombinant human or humanized antibodies.
* Presence of any psychological, familial, sociological, or geographical condition potentially hampering compliance with the study protocol and follow-up schedule; those conditions should be discussed with the patient before registration in the trial.
* Participation in another clinical study (except sub studies of this protocol) within the 30 days before randomization and during this study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2013-06; Primary Completion 2016-09 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
Progression free survival | 1 year
  Increase in progression free survival rate at 1 year in each experimental arm (mFOLFOX6 + bevacizumab or panitumumab) compared to mFOLFOX6 alone arm.

SECONDARY OUTCOMES:
Pathological response rate | 4 years
  Increase in major pathological response rate between mFOLFOX6 alone arm and each experimental arm.
Resection rate | 4 years
  Compare the percentage of patients with total resection with these three treatments.
Overall survival | 8 years
  Overall survival is defined as the time interval between the date of randomization and the date of death. Patients who are still alive when last traced will be censored at the date of last follow-up.
Safety | 4 years
  All adverse events will be recorded; the investigator will assess whether those events are drug related (reasonable possibility, no reasonable possibility) and this assessment will be recorded in the database for all adverse events.

CONTACTS AND LOCATIONS:
Overall Officials: Bernard Nordlinger, Pr., Study Chair — C.H.U. AMBROISE PARE AP-HP, Boulogne-Billancourt, France; Stephane Benoist, Pr., Study Chair — HOPITAL DE BICETRE AP-HP, Le Kremlin Bicetre, France
Locations (25):
- Allgemeines Krankenhaus der Stadt Wien, Vienna, Austria
- Belgium (5):
  - Hopital Universitaire Brugmann, Brussels
  - Universitair Ziekenhuis Gent, Ghent
  - AZ Groeninge Kortrijk - Campus Kennedylaan, Kortrijk
  - AZ Turnhout - Campus Sint Elisabeth, Turnhout
  - Centre Hospitalier Peltzer-La Tourelle, Verviers
- France (16):
  - Institut Sainte Catherine, Avignon
  - Institut Bergonie, Bordeaux
  - CHU Ambroise Pare, Boulogne-Billancourt
  - Assistance Publique - Hôpitaux de Paris - Hopital De Bicetre AP-HP, Le Kremlin-Bicêtre
  - Centre Hospitalier Saint Joseph Saint Luc, Lyon
  - Centre Leon Berard, Lyon
  - Hopital Prive Jean Mermoz, Lyon
  - Centre Antoine Lacassagne, Nice
  - Hopital Europeen Georges Pompidou, Paris
  - Groupe Hospitalier Diaconesses Croix Saint-Simon - Site Reuilly, Paris
  - CHU de Lyon - Centre Hospitalier Lyon Sud, Pierre-Benite (lyon)
  - CHU de Reims - Hôpital Robert Debré, Reims
  - Hopital Charles Nicolle, Rouen
  - Centre Hospitalier Privé Saint-Grégoire, Saint-Grégoire
  - CHU Saint-Etienne - CHU de Saint-Etienne - Hopital Nord, Saint-Priest-en-Jarez
  - CHU d'Amiens - CHU Amiens - Hopital Sud, Salouël
- The Netherlands Cancer Institute-Antoni Van Leeuwenhoekziekenhuis, Amsterdam, Netherlands
- Hospital General Vall D'Hebron, Barcelona, Spain
- Hôpitaux universitaires de Genève - HUG - site de Cluse-Roseraie, Geneva, Switzerland